CLINICAL TRIAL: NCT01693471
Title: Survey on the Effect of Health Related QOL Associated With Compliance of Carbocisteine in Asthma Patients Study (SEARCH Study)
Brief Title: Survey on the Effect of Health Related Quality of Life (QOL) Associated With Compliance of Carbocisteine in Asthma Patients
Status: Completed | Type: Observational
Sponsor: Kyorin Pharmaceutical Co.,Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: SEARCH-2012
Record Dates: First submitted 2012-09-21; First posted 2012-09-26 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-02

CONDITIONS: Asthma
Keywords: asthma; SF-36; HRQOL
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SEARCH Study Group

SUMMARY:
The objectives of this study are to investigate the influence on HR-QOL (SF-36 v2) resulting from the compliance of MUCODYNE Tablets or MUCODYNE DS (Dry Syrup) 50% in asthma patients whose control levels are partly controlled or uncontrolled.

DETAILED DESCRIPTION:
Period: 2012-2013 Observation Time: 0 week, 4 week

Matters investigated:

1. QOL determination using SF-36 v2
2. Medication compliance (VAS scale)
3. Gender, age, diagnosis, asthma subtype, severity, duration of disease, level of asthma control, concomitant drugs, comorbidities, smoking, alcohol, work

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥ 20 years of age
* Outpatients
* Patients with mild or moderate persistent asthma
* Patients with phlegm
* Patients whose levels of asthma control are partly controlled or uncontrolled
* Patients who are planned to treat MUCODYNE
* Patients who voluntarily submitted written consent forms upon participation in this study

Exclusion Criteria:

* Patients with a history of adverse reactions to carbocisteine
* Patients with serious cardiac, hepatic, renal, pulmonary, or hematological disease
* Patients with the possibility of pregnancy or suspected pregnancy
* Patients with complication of malignancy
* Current smoker
* Patients with definitive diagnosis for COPD
* Other patients whom investigators or subinvestigators considered inappropriate to participate in this study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General Practitioner
Sampling Method: Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Score of SF-36 | 4 week

SECONDARY OUTCOMES:
HR-QOL condition of asthma patients with phlegm | 0 week
Medication compliance: measured by patient response to visual analog scale | 4 week
Relation between a medication compliance measured by patient response to visual analog scale and change of HR-QOL from baseline at 4 weeks | 0 week, 4 week

CONTACTS AND LOCATIONS:
Overall Officials: Akito Saegusa, Mr., Study Chair — Kyorin Pharmaceutical Co.,Ltd
Locations (1):
- Senzoku Respiratory Disease and Allergy Clinic, Ōta-ku, Tokyo, Japan